CLINICAL TRIAL: NCT02030262
Title: Study of the Impact of Air Versus SF6 20% on Visual Acuity Improvement After Epiretinal Membrane Stripping
Brief Title: Study of Impact of Air vs SF6 20% on Visual Acuity Improvement After Epiretinal Membrane Stripping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C13-10-1231
Record Dates: First submitted 2014-01-07; First posted 2014-01-08 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Epiretinal Membrane
MeSH Terms: conditions — Epiretinal Membrane

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Air (Experimental): The participant will undergo epiretinal membrane peeling with fluid-air exchange. The remaining of the surgery is the same in all arms.
  Interventions: Procedure: Epiretinal membrane peeling with fluid-air exchange
- Sulfur hexafluoride (SF6) (Active Comparator): The participant will undergo epiretinal membrane peeling with fluid-SF6 exchange. The remaining of the surgery will stay the same.
  Interventions: Procedure: Epiretinal membrane peeling with fluid-SF6 exchange

INTERVENTIONS:
Procedure: Epiretinal membrane peeling with fluid-air exchange — The intervention starts with a pars plana vitrectomy and then a epiretinal membrane peeling is performed. During the fluid-gaz exchange, the gaz used will be air. The remaining of the intervention is the same between the two arms.
  Arms: Air
Procedure: Epiretinal membrane peeling with fluid-SF6 exchange — The intervention starts with a pars plana vitrectomy and then a epiretinal membrane peeling is performed. During the fluid-gaz exchange, the gaz used will be SF6 (sulfur hexafluoride). The remaining of the intervention is the same between the two arms.
  Arms: Sulfur hexafluoride (SF6)

SUMMARY:
The purpose of this study is to determine if one of these gaz (air and sulfur hexafluoride) is better than the other in epiretinal membrane peeling surgery. Both are already used for this surgery and this study will tell us if one is better than the other.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of epiretinal membrane with corresponding optical coherence tomography
* ETDRS visual acuity worse or equal to 20/30
* Adult able to give consent

Exclusion Criteria:

* Diagnosis of age-related macular degeneration
* Opacity blocking the fundus visualisation
* Presence of active intraocular inflammation
* Presence of intraocular tumor
* Presence of retinal detachment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-12; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Visual acuity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu Caissie, MD, FRCSC, Principal Investigator — Centre de recherche du CHU de Québec; Université Laval
Locations (1):
- Centre universitaire d'ophtalmologie, Hôpital du Saint-Sacrement, CHU de Québec, Québec, Quebec, Canada